CLINICAL TRIAL: NCT02081209
Title: Non-Invasive Fat Layer Reduction in the Lateral Thighs With a Cryolipolysis System Using Varied Treatment Parameters
Brief Title: Outer Thigh Study With Varied Treatment Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA14-001
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction

STUDY DESIGN:
Intervention Model Description: All subjects to be treated on one lateral thigh at a protocol-defined temperature for 120 minutes. Treatment of the contralateral thigh was performed using two unique protocol-defined temperatures for 60 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lateral Thigh Treatment Group (Experimental): All subjects were treated on both thighs with the CoolSculpting System. One lateral thigh was treated using a protocol-defined temperature for 120 minutes. The contralateral thigh was treated at a protocol defined temperature for 60 minutes for 18 subjects. Twenty-two subjects were treated on the contralateral outer thigh with a 3rd protocol-defined temperature for 60 minutes.
  Interventions: Device: The Zeltiq CoolSculpting System

INTERVENTIONS:
Device: The Zeltiq CoolSculpting System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis

SUMMARY:
The purpose of this study is to compare the performance of the Zeltiq CoolSculpting System using various treatment parameters for non-invasive reduction of subcutaneous fat in the lateral thighs.

DETAILED DESCRIPTION:
The purpose of this study is to compare the performance of a cryolipolysis system using various treatment parameters for non-invasive reduction of subcutaneous fat in the lateral thighs.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects > 18 years of age and < 65 years of age.
2. Subject has clearly visible fat on the intended treatment area (lateral thighs), which in the investigator's opinion, may benefit from the treatment.
3. Subject has not had weight change exceeding 10 pounds in the preceding month.
4. Subject with body mass index (BMI) up to 30. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
5. Subject agrees to maintain his/her weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
6. Subject has read and signed a written informed consent form.

Exclusion Criteria

1. Subject has had a surgical procedure(s) in the area of intended treatment.
2. Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
3. Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 2 months.
4. Subject has significant asymmetry between the lateral thighs.
5. Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
6. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
7. Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
8. Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
9. Subject is taking or has taken diet pills or supplements within the past month.
10. Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
11. Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
12. Subject is pregnant or intending to become pregnant during the study period (in the next 5 months).
13. Subject is lactating or has been lactating in the past 6 months.
14. Subject is unable or unwilling to comply with the study requirements.
15. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
16. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2014-10-21 (Actual); Study Completion 2014-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bachelor, MD, Principal Investigator — Innovation Research Center
Locations (2):
- United States (2):
  - Marina Plastic Surgery, Marina del Rey, California
  - Innovation Research Center, Pleasanton, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 40 enrolled subjects, initiated treatment and had safety evaluations after treatment (safety population). The Per-Protocol Population included all treated subjects who completed treatment, were followed for 16 weeks and who did not become pregnant and with weight change of no more than 5 pounds at the time the final post-treatment images were taken.
Groups:
- Lateral Thigh Treatment Group: Each subject was treated on one lateral thigh at -10 degrees C. The contralateral thigh was treated at -13 degrees C for 60 minutes for 18 subjects. The contralateral thigh on 21 subjects was treated at -15 degrees for 60 minutes.
Period: Overall Study
Arm/Group | Lateral Thigh Treatment Group
Started | 40 (All subjects treated on one lateral thigh at -10 C; contralateral thigh was treated using -13 C or -15 C.)
Initiated -10C and -13C Treatment | 18
Initiated -10C and -15C Treatment | 22
Completed -10C and -13C Treatment | 18
Completed -10C and -15C Treatment | 21 (One subject received an incomplete treatment, therefore 39 subjects are included in the as-treated population.)
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Lateral Thigh Treatment Group: Non-invasive fat reduction of both lateral thighs was performed using the Zeltiq CoolSculpting System.
Arm/Group | Lateral Thigh Treatment Group
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 43.0 [27 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1
  Asian | 1
  Hispanic | 5
  Caucasian | 31
  Others | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Body Mass Index [Mean (Full Range); unit: kg//m^2] | 24.4 [19.2 to 29.6]

OUTCOME MEASURES:

1. Primary Outcome: Safety of the Zeltiq Device
Description: The number of device- or procedure-related adverse events will be tabulated from the time of enrollment through the 16 week follow-up visit.
Time Frame: Time of enrollment though16 weeks post-treatment (approximately 5 months)
Population: All subjects treated with the Zeltiq CoolSculpting System were included in the analysis population.
Measure: Number; unit: device/procedure related AEs
Groups:
- Lateral Thigh Treatment Parameter: -10C: All subjects received treatment on one (1) lateral thigh at -10C.
- Contralateral Thigh Treatment Parameter: -13C: Subjects with contralateral lateral thigh treatment at -13C.
- Contralateral Thigh Treatment Parameter:-15C: Contralateral lateral thigh was treated using -15C.
Arm/Group | Lateral Thigh Treatment Parameter: -10C | Contralateral Thigh Treatment Parameter: -13C | Contralateral Thigh Treatment Parameter:-15C
Number analyzed (Participants) | 40 | 18 | 22
device/procedure related AEs | 7 | 4 | 12

2. Primary Outcome: Safety of the Zeltiq Device
Description: The number of unanticipated adverse device effects (UADEs) will be tabulated.
Time Frame: From enrollment through 16 week follow-up (approximately 5 months)
Population: All subjects treated with the Zeltiq CoolSculpting System were included in the analysis population.
Measure: Number; unit: UADEs reported
Groups:
- Contralateral Thigh Treatment Parameter: -13C: Contralateral lateral thigh treated at -13C.
Arm/Group | Lateral Thigh Treatment Parameter: -10C | Contralateral Thigh Treatment Parameter: -13C | Contralateral Thigh Treatment Parameter:-15C
Number analyzed (Participants) | 40 | 18 | 22
UADEs reported | 0 | 0 | 0

3. Primary Outcome: Percentage of Pre-treatment Images Correctly Identified.
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Criteria for evaluable photos for the purposes of the independent review: subject completed treatment regimen; subject has complete set of baseline photos; subject has a complete set of post-treatment photos; photos were taken using Zeltiq standard procedure. The expected success rate is 80%.
Time Frame: Baseline and 16 weeks post-treatment
Population: The per-protocol analysis population included subjects with available photos and complied with protocol-defined weight maintenance. Thirty-four subjects had 68 photo pairs which were presented to three blinded physician reviewers.Of the 37 subjects with available photos, 3 subjects were excluded due to weight change outside of protocol requirements.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Groups:
- All Subjects Both Outer Thighs: All subjects with evaluable images from both outer thighs are included.
- Lateral Thigh Treatment Group-All Subjects: Non-invasive fat reduction of lateral thighs was performed using the Zeltiq CoolSculpting System. Each subject in the treatment group had one lateral thigh treated with uniform treatment parameters (Treatment type 1).
- Group 1: Contralateral Outer Thigh Treatment 2: Each subject in the group received treatment type 2 on the contralateral outer thigh.
- Contralateral Outer Thigh Treatment Group 3: Each subject in the group received treatment with Type 3 treatment parameters on the contralateral outer thigh.
Arm/Group | All Subjects Both Outer Thighs | Lateral Thigh Treatment Group-All Subjects | Group 1: Contralateral Outer Thigh Treatment 2 | Contralateral Outer Thigh Treatment Group 3
Number analyzed (Participants) | 34 | 34 | 16 | 18
Number analyzed (photos) | 204 | 102 | 48 | 54
photos | 168 | 79 | 38 | 51
Statistical Analysis 1: Comparison: All Subjects Both Outer Thighs; Test type: Other; sucess percentage = 82.4, 95% CI 2-sided [76.4 to 87.3]
Statistical Analysis 2: Comparison: Lateral Thigh Treatment Group-All Subjects; Test type: Other; sucess percentage = 77.4, 95% CI 2-sided [68.1 to 85.1]
Statistical Analysis 3: Comparison: Group 1: Contralateral Outer Thigh Treatment 2; Test type: Other; sucess percentage = 79.2, 95% CI 2-sided [65.0 to 89.5]
Statistical Analysis 4: Comparison: Contralateral Outer Thigh Treatment Group 3; Test type: Other; sucess percentage = 94, 95% CI 2-sided [84.6 to 98.8]

4. Secondary Outcome: Change in the Fat Layer of the Treated Area as Measured by Ultrasound
Description: Change in the fat layer thickness will be calculated by comparison of pre-treatment and 16 week post-treatment ultrasound measurements taken in the area treated with the device, and in the adjacent untreated control area. The Sponsor's standardized techniques for obtaining ultrasound imaging will be used. Overall fat layer thickness changes were normalized for each subject by subtracting the change in control (untreated area) from the change in treated area to remove the influence of weight variations. Success is defined as, on average, at least a 1mm or greater reduction in fat layer thickness for the treated region as compared to the untreated control. Results indicate the mean fat layer reduction in mm.
Time Frame: 16 weeks post-treatment
Population: The per-protocol analysis population included 33 subjects with available ultrasound images for both lateral thighs, resulting in 66 images for analysis.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Group 1: All Subjects First Outer Thigh Treatment: Treatment type 1 was administered to all subjects in Group 1.
- Contralateral Thigh Treatment Group 2: All subjects received treatment type 2 on the contralateral thigh.
- Contralateral Thigh Treatment Group 3: All subjects received treatment type 3 on the contralateral thigh.
Arm/Group | Group 1: All Subjects First Outer Thigh Treatment | Contralateral Thigh Treatment Group 2 | Contralateral Thigh Treatment Group 3
Number analyzed (Participants) | 33 | 15 | 18
mm | -2.3 (1.9) | -1.3 (1.5) | -3.0 (2.2)
Statistical Analysis 1: Comparison: Group 1: All Subjects First Outer Thigh Treatment; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 2.3, Standard Deviation 1.9
Statistical Analysis 2: Comparison: Contralateral Thigh Treatment Group 2; Test type: Other; Mean Difference (Net) = 1.3, 95% CI 2-sided [0.5 to 2.1]
Statistical Analysis 3: Comparison: Contralateral Thigh Treatment Group 3; Test type: Other; Mean Difference (Net) = 3.0, 95% CI 2-sided [2.0 to 4.1]

5. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction with the Zeltiq procedure as determined by the results of a subjects satisfaction questionnaire at the 16 week follow up visit. The questionnaire is composed of a 5-point Likert scale questions, as well as free text responses. Subjects will be asked to determine overall satisfaction with the treatment. The choices will be 1) very unsatisfied; 2) somewhat unsatisfied; 3) neither unsatisfied or satisfied; 4) somewhat satisfied; 5) very satisfied.
Time Frame: 16-weeks post treatment
Population: Subjects completing the questionnaire at the 16-week follow-up visit were included in the analysis population.
Measure: Count of Participants; unit: Participants
Groups:
- CoolSculpting of the Lateral Thigh Group: Non-invasive fat reduction of both lateral thighs was performed using the Zeltiq CoolSculpting System.
Arm/Group | CoolSculpting of the Lateral Thigh Group
Number analyzed (Participants) | 38
Participants
  Procedure very to somewhat comfortable | 22
  Very to somewhat comfortable during weeks post procedure | 25
  Very visible to somewhat visible fat reduction | 36
  More than or about expected overall effect | 28
  Very to somewhat satisfied with procedure | 32
Statistical Analysis 1: Comparison: CoolSculpting of the Lateral Thigh Group; Test type: Other; Data from the 16-week follow-up questionnaire were tabulated for all subjects with completed questionnaires.. All confidence intervals were calculated at 95%. Alpha was calculated to be 0.05, critical probability (p*) was calculated to be 0.975. Assuming normal distribution of survey recipients, a standard deviation of 1.96 is used to calculate the standard margin of error

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment through the 16-week follow-up visit, approximately 5 months.
Description: The Safety Population consists of all enrolled participants who received a treatment session (started or completed).
  AEs of Nausea, Seasonal Allergies, Sinus Cold, Lumbar Cyst, Surgical Procedure, Menstrual Irregularity, Uterine Fibroid, and Pneumonia are presented in multiple arms because they were not attributable to a given intervention.
  One incident of Prolonged Sensory Alteration Post Procedure that occurred outside of the treatment area was reported for -10 C and -15 C arms.
Arm/Group | Lateral Thigh Treatment Parameter: -10C | Contralateral Thigh Treatment Parameter: -13C | Contralateral Thigh Treatment Parameter:-15C
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 17/40 | 6/18 | 20/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lateral Thigh Treatment Parameter: -10C (N=40) | Contralateral Thigh Treatment Parameter: -13C (N=18) | Contralateral Thigh Treatment Parameter:-15C (N=22)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Prolonged sensory alteration post procedure (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4) | 4 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus cold (General disorders) | 2 (2) | 0 (0) | 2 (2)
Uterine fibroid (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Menstrual irregularity (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical procedure (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Lumbar cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Seasonal allergies (General disorders) | 1 (1) | 0 (0) | 1 (1)
Dry, flaky skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No